CLINICAL TRIAL: NCT03144921
Title: EPIC: A Group-based Intervention for Early-stage AD Dyads in Diverse Communities
Brief Title: EPIC: An Intervention for Early-stage AD Dyads - Adapted for Virtual Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, David W Coon, Associate Dean, R.I.S.E. and Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005510, STUDY00012907
Record Dates: First submitted 2017-05-02; First posted 2017-05-09 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Dementia; Alzheimer Disease; Memory Loss
Keywords: Early-stage Dementia; Early-stage Alzheimer's disease; Care partner; Caregivers; Caregiving
MeSH Terms: conditions — Dementia; Alzheimer Disease; Memory Disorders

STUDY DESIGN:
Intervention Model Description: Dyads will be randomized (assigned by chance) to one of two groups: 10 EPIC A or 2) EPIC B (Wait List Control - WLC. Randomization with stratification by language preference (English vs. Spanish) and geographic setting will occur in sets of 4 to 8 (average 6) eligible dyads.
  The RCT ends at T2 with comparison of changes in outcomes between EPIC and WLC participants from Assessment 1 (baseline) to Assessment 2 (3 months post baseline). T2-T3 assessments will be used for within-group and maintenance of gains analyses from about 3 months to 6 months post baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EPIC A (Experimental): Group A will start the EPIC intervention immediately after assessment 1. The EPIC program consists of a 7-session, psychoeducational skills training intervention, held via Zoom, designed to provide education and skills on how to prepare for the future and reduce stress regarding memory changes and loss for both the person with early-stage dementia and their care partner. Following the 7 EPIC sessions, participants will attend monthly booster sessions, held via Zoom, to reinforce the skills/lessons. Participants may voluntarily choose to continue attending booster sessions through 2024.
  Interventions: Behavioral: psychoeducational skills training intervention
- EPIC B (WLC) (Active Comparator): Group B - the wait list comparison (WLC) group - will have a 75-minute group education session (comparator intervention), held via Zoom, about 3 weeks after baseline assessment. The WLC session is an overview of memory loss/dementia and its related impact for EPs and CPs and an overview of aging network services in the community. They will receive a brief telephone check-in call approximately 3 weeks before the T2 assessment. The WLC group will start the complete EPIC psychoeducational skills training intervention, held via Zoom, immediately after Assessment 2. Following completion of the 7 EPIC sessions, participants will attend monthly booster sessions, held via Zoom, to reinforce the skills/lessons. Participants may voluntarily choose to continue attending booster sessions through 2024.
  Interventions: Behavioral: psychoeducational skills training intervention

INTERVENTIONS:
Behavioral: psychoeducational skills training intervention — This protocol is a minimal risk care values clarification /care planning and psychoeducational skills training intervention, delivered as a workshop series plus one in-home session for people in the early stages of memory loss and their care partner together.

SUMMARY:
EPIC II (Early-Stage Partners in Care) is a research project designed to assist people with early-stage memory loss and their care partners by providing early-stage related education and skill-training sessions, held via Zoom, designed to reduce stress, enhance well-being, manage challenges, and plan for the future. Researchers will gather feedback from individuals about their experience to continue to improve programs for early-stage memory loss.

DETAILED DESCRIPTION:
The purpose of this study is to help early-stage individuals who have early-stage memory loss or early stage dementia and their current or future care partners by providing education and skill-training programs, held via Zoom, designed to reduce stress and distress, increase well-being and quality of life, and plan for the future. About 160 early-stage dyads (person with early-stage dementia and his/her care partner) will be enrolled across the United States through Arizona State University.

People who decide to voluntarily participate in this program, will be asked to:

* Meet others with memory loss and their care partners.
* Attend six group sessions via Zoom (2 hours & 30 minutes each) to learn strategies to help handle new situations, reduce stress, improve mood, communicate better with each other, and plan for the future.
* Participate in one 90-minute individualized session via Zoom to address specific issues that may be unique to each dyad's situation.
* Participate in three 2-hour confidential interviews that involve questions about background, mood, and quality of life.
* Participate in interviews at the start, and again about 3 and 6 months, via Zoom, to help us to continue to improve the program.
* Attend several monthly booster sessions after completion of the seven EPIC sessions.

Each person will receive up to $45 for completing all follow-up interviews, or $20- 25 for each interview completed. All participants are offered the EPIC sessions shortly after their first interview or shortly after their 3-month interview. Some participants will also attend an additional free education workshop within one month of the initial assessment.

ELIGIBILITY:
DYAD INCLUSION CRITERIA:

1. All participants - Care Partners (CP) and Early-Stage People (EP) - will be at least 18 years of age and speak, read, and write English or Spanish.
2. Eligible dyad relationships include spouse, adult-child relationships (e.g., daughters), and other close friends and family members.
3. Care partners must self-identify as the person who currently has or who expects to have the most hands-on responsibility and ongoing involvement with the EP.
4. CPs must live with or have regular contact with the EP.
5. EPs and CPs must reside in a community setting.

EP INCLUSION CRITERIA:

1. Live at home rather than an institutional setting,
2. Have a confirmed diagnosis of OR symptoms consistent with early-stage dementia
3. Exhibit changes in memory as specified on the AD8 dementia screening tool.
4. Have a Mini-Mental State Exam (MMSE)i score within a protocol-specified range.
5. Have a CP who is defined by the EP as being the unpaid "family member" who has or will have primary responsibility for providing assistance to the EP

EP EXCLUSION CRITERIA:

1. Denying or not reporting any trouble with memory, based on self-report
2. Normal cognition, based on score derived from screening tool
3. If yes to BOTH:

   1. severe mental illness or developmental disability before the age of 45
   2. memory problems due to past head injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
EP and CP Emotional well-being | Assessments T1-T3 to be conducted over span of six months
  Examine the efficacy of the EPIC intervention as compared with a Wait List Comparison condition by looking at the change over time in the Positive and Negative Affect Scales (Dementia Quality of Life Instrument).
EP Quality of Life | Assessments T1-T3 to be conducted over span of six months
  Assess EP Quality of life and CPs perception of EPs Quality of life by looking at the change over time in the Quality of Life Measure in Dementia.

SECONDARY OUTCOMES:
Knowledge and Use of Services for People with Dementia and their Care Partners | Assessments T1-T3 to be conducted over span of six months
  Assess the knowledge of, use of, and satisfaction with a variety of services (for example, respite, support groups, case management, referral services) relevant to people with dementia and their care partners by looking at the change over time.
Communication Skills and Support within the Dyad | Assessments T1-T3 to be conducted over span of six months
  Assess communication by looking at the change over time in the Dyadic Relationship Scale and Emotional Intimacy Disruptive Behavior Scale.
EP and CP Care preparedness | Assessments T1-T3 to be conducted over span of six months
  Assess EP and CP perceptions of how well prepared they feel for addressing future care needs by looking at the change over time in the Care Partners Preparedness Scale (modified).

OTHER OUTCOMES:
Initial incremental cost effectiveness of EPIC compared with Wait List Comparison condition | T1 - T2 Assessments (Baseline to 3 months)
  Based on Quality of Life Adjusted Years for the EPs and hours providing care for CPs, conduct a cost benefit analysis to explicitly indicate whether benefits of the EPIC program outweigh costs by looking at the change over time.

CONTACTS AND LOCATIONS:
Overall Officials: David W. Coon, PhD, Principal Investigator — Arizona State University
Locations (1):
- Nationwide Program Locations (Based at ASU Edson College of Nursing and Health Innovation), Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No